CLINICAL TRIAL: NCT01811212
Title: Phase II Study of Cabozantinib in Patients With Radioiodine-Refractory Differentiated Thyroid Cancer Who Progressed on Prior VEGFR-Targeted Therapy
Brief Title: Cabozantinib-S-Malate in Treating Patients With Refractory Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00554; NCI-2013-00554 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012C0101; RU241210I; OSU 12154; 9312 (Other: Ohio State University Comprehensive Cancer Center); 9312 (Other: CTEP); N01CM00039 (NIH); N01CM00070 (NIH); N01CM00071 (NIH); N01CM00099 (NIH); P30CA016058 (NIH); UM1CA186705 (NIH)
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Results first posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Poorly Differentiated Thyroid Gland Carcinoma; Recurrent Thyroid Gland Carcinoma; Stage I Thyroid Gland Follicular Carcinoma; Stage I Thyroid Gland Papillary Carcinoma; Stage II Thyroid Gland Follicular Carcinoma; Stage II Thyroid Gland Papillary Carcinoma; Stage III Thyroid Gland Follicular Carcinoma; Stage III Thyroid Gland Papillary Carcinoma; Stage IVA Thyroid Gland Follicular Carcinoma; Stage IVA Thyroid Gland Papillary Carcinoma; Stage IVB Thyroid Gland Follicular Carcinoma; Stage IVB Thyroid Gland Papillary Carcinoma; Stage IVC Thyroid Gland Follicular Carcinoma; Stage IVC Thyroid Gland Papillary Carcinoma; Tall Cell Variant Thyroid Gland Papillary Carcinoma; Thyroid Gland Oncocytic Follicular Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary; Thyroid cancer, Hurthle cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cabozantinib-s-malate) (Experimental): Patients receive cabozantinib-s-malate PO daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib S-malate; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Cabozantinib S-malate — Given PO
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well cabozantinib-s-malate works in treating patients with thyroid cancer that does not respond to treatment. Cabozantinib-s-malate may stop the growth of thyroid cancer by blocking some of the enzymes needed for cell growth. Cabozantinib-s-malate may also stop the growth of thyroid cancer by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The objective response rate, defined as the proportion of patients who have had a partial response (PR) or complete response (CR) within the first 6 months after initiation of therapy with cabozantinib (cabozantinib-s-malate).

SECONDARY OBJECTIVES:

I. To assess duration of objective response, progression-free survival and overall survival.

II. To assess tolerability and adverse events of cabozantinib as a 2nd line therapy in patients with differentiated thyroid cancer (DTC).

TERTIARY OBJECTIVES:

I. To assess effect of cabozantinib on serum tumor marker thyroglobulin and its correlation with overall response rate.

II. To assess response of cabozantinib in bone metastasis (bone metastasis-specific progression free survival) as evaluated by pre- and on-study functional imaging such as bone scan, fludeoxyglucose F 18 (18F-FDG) positron emission tomography (PET) scan and/or 18F sodium fluoride (NaF) PET scan.

III. To assess effect of cabozantinib on serum and urinary markers of bone turnover and its correlation with response to bone metastasis.

IV. To assess predictors of response by performing tumor genotype studies (e.g. v-raf murine sarcoma viral oncogene homolog B [BRAF], rat sarcoma [RAS], phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha [PIK3CA], mitogen-activated protein kinase 1 [MAP2K1], v-akt murine thymoma viral oncogene homolog 1 [AKT1], mesenchymal-epithelial transition [MET], rearranged in transformation [RET]/papillary thyroid carcinoma [PTC] rearrangement) in archived tumor tissue.

V. To assess predictors of response by assessing baseline expression levels of vascular endothelial growth factor (VEGF), phosphorylated vascular endothelial growth factor receptor (pVEGFR), phosphorylated mitogen-activated protein kinase 1 (pERK), phosphorylated AKT1 (pAKT) and/or total met proto-oncogene (MET) by immunohistochemistry in archived tumor tissue.

OUTLINE:

Patients receive cabozantinib-s-malate orally (PO) daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks and then every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed papillary thyroid cancer, follicular thyroid cancer or hurthle cell thyroid cancer (cancer, follicular variant of papillary thyroid cancers or any of the above mixed histology will be allowed; these patients will be enrolled on Arm A of the trial); patients with the following aggressive histologies will be enrolled on Arm B of the trial; tall cell, insular or poorly differentiated thyroid cancer
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 2.0 cm with conventional techniques or as >= 1.0 cm (or >= 1.5 cm in short axis for lymph node) with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Patients must have radioactive iodine (RAI)-refractory/resistant disease as defined by one or more of the following criteria:

  * One or more measurable lesions that do not demonstrate RAI uptake
  * One or more measurable lesions progressive by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 within 12 months of prior RAI therapy
  * One or more measurable lesion present after cumulative RAI dose of >= 600 mCi
* Patients must have "progressed on" up to 2 lines of prior vascular endothelial growth factor receptor (VEGFR)-targeted therapy (including but not limited to sorafenib, sunitinib, vandetanib, pazopanib, or lenvatinib) as defined by progressive disease per RECIST while receiving VEGFR-targeted therapy; Note: patients who progressed on kinase inhibitor that target VEGFR and MET will not be eligible
* Prior external beam radiation, systemic cytotoxic chemotherapy or BRAF- or non-VEGFR-targeted therapies will be allowed, provided that >= 4 weeks has elapsed since receiving prior treatment and they have recovered to =< grade 1 treatment-related toxicities
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil count >= 1,500/mcL
* Platelet count >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Thyroid stimulating hormone (TSH) < lower limit of normal (LLN) (patients not able to tolerate TSH suppression can be granted an exception)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (patients [Pts] with Gilbert's syndrome are excluded from this requirement)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3.0 x institutional upper limit of normal
* Creatinine =< 1.5 x ULN
* Serum albumin >= 2.8 g/dL
* Lipase < 2.0 x ULN and no radiologic or clinical evidence of pancreatitis
* Urine protein/creatinine ratio (UPCR) =< 1
* Serum phosphorus, calcium, magnesium and potassium >= LLN
* Prothrombin time (PT) < 1.3 x ULN
* International normalized ratio (INR) < 1.3 x ULN
* Partial thromboplastin time (PTT) test < 1.3 x ULN
* Women of childbearing potential must have a negative pregnancy test at screening; women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal; postmenopause is defined as amenorrhea >= 12 consecutive months; Note: women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, ovarian suppression or any other reversible reason
* Women of child-bearing potential and men must agree to use adequate contraception; women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of cabozantinib administration; sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used; all subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 4 months after the last dose of study drug(s)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior treatment with cabozantinib or any tyrosine kinase inhibitor that targets MET or monoclonal antibody (mAb) targeting MET (such as onartuzumab [MetMAb])
* The subject has received radionuclide treatment =< 6 weeks of the first dose of study treatment
* The subject has received any other type of investigational agent =< 28 days before the first dose of study treatment
* The subject has not recovered to baseline or Common Terminology Criteria for Adverse Events (CTCAE) =< grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant adverse events (AEs)
* The subject has active brain metastases or epidural disease; subjects with brain metastases previously treated with whole brain radiation or radiosurgery or subjects with epidural disease previously treated with radiation or surgery who are asymptomatic and do not require steroid treatment for at least 2 weeks before starting study treatment are eligible; baseline brain imaging with contrast-enhanced CT or MRI scans for subjects with known brain metastases is required to confirm eligibility; eligible patients with brain metastases can be taking anti-convulsant medications but only non-enzyme inducing anti-epileptic agents (NEIAED) will be allowed
* The subject requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or factor xabans (Xa) inhibitors, or antiplatelet agents (e.g., clopidogrel); low dose aspirin (=< 81 mg/day), low-dose warfarin (=< 1 mg/day), and prophylactic low molecular weight heparin (LMWH) are permitted
* The subject requires chronic concomitant treatment of strong cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St. John's Wort) or strong CYP3A4 inhibitors (ketoconazole, itraconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, voriconazole, and posaconazole); Note: because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated lists; medical reference texts such as the Physicians' Desk Reference may also provide this information; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* The subject has experienced any of the following:

  * Clinically-significant gastrointestinal bleeding =< 6 months before the first dose of study treatment
  * Hemoptysis of >= 0.5 teaspoon (2.5 mL) of red blood =< 3 months before the first dose of study treatment
  * Any other signs indicative of pulmonary hemorrhage =< 3 months before the first dose of study treatment
* The subject has radiographic evidence of cavitating pulmonary lesion(s)
* The subject has tumor that is invading or encasing any major blood vessels
* The subject has evidence of tumor invading the gastrointestinal (GI) tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor =< 28 days before the first dose of cabozantinib
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders including:

    * Congestive heart failure (CHF): New York Heart Association (NYHA) class III (moderate) or class IV (severe) at the time of screening
    * Concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mmHg systolic, or > 90 mmHg diastolic despite optimal antihypertensive treatment =< 7 days of the first dose of study treatment
    * Any history of congenital long QT syndrome
    * Any of the following =< 6 months before the first dose of study treatment:

      * Unstable angina pectoris
      * Clinically-significant cardiac arrhythmias
      * Stroke (including transient ischemic attack [TIA], or other ischemic event)
      * Myocardial infarction
      * Thromboembolic event requiring therapeutic anticoagulation (Note: subjects with a venous filter [e.g. vena cava filter] are not eligible for this study)
  * Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including:

    * Any of the following =< 28 days before the first dose of study treatment

      * Intra-abdominal tumor/metastases invading GI mucosa
      * Active peptic ulcer disease as evidenced by esophagogastroduodenoscopy (EGD)
      * Inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
      * Malabsorption syndrome
    * Any of the following =< 6 months before the first dose of study treatment:

      * Abdominal fistula
      * Gastrointestinal perforation
      * Bowel obstruction or gastric outlet obstruction
      * Intra-abdominal abscess; Note: complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more than 6 months before the first dose of study treatment
  * Other disorders associated with a high risk of fistula formation including percutaneous endoscopic gastrostomy (PEG) tube placement =< 3 months before the first dose of study therapy
  * Other clinically significant disorders such as:

    * Active infection requiring systemic treatment =< 28 days before the first dose of study treatment
    * Serious non-healing wound/ulcer/bone fracture =< 28 days before the first dose of study treatment
    * History of organ transplant
    * History of major surgery as follows:

      * Major surgery =< 3 months of the first dose of cabozantinib if there were no wound healing complications or =< 6 months of the first dose of cabozantinib if there were wound complications
      * Minor surgery =< 1 months of the first dose of cabozantinib if there were no wound healing complications or =< 3 months of the first dose of cabozantinib if there were wound complications
      * In addition, complete wound healing from prior surgery must be confirmed at least 28 days before the first dose of cabozantinib irrespective of the time from surgery
* The subject is unable to swallow tablets
* The subject has a corrected QT interval calculated by the Fridericia or Bazett's formula (QTcF) > 480 ms within 28 days before registration; Note: if initial QTcF or QTcB is found to be > 480 ms, two additional electrocardiograms (EKGs) separated by at least 3 minutes should be performed; if the average of these three consecutive results for QTcF or QTcB is =< 480 ms, the subject meets eligibility in this regard
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee
* The subject has had evidence within 2 years of the start of study treatment of another malignancy which required systemic treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cabozantinib
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy; Note: patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* The subject has received prior treatment with a small molecule kinase inhibitor or a hormonal therapy (including investigation kinase inhibitors or hormones) within 14 days or five half-lives of the compound or active metabolites, whichever is longer, before the first dose of the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-05-08 (Actual); Primary Completion 2015-07-13 (Actual); Study Completion 2017-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Shah, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (7):
- United States (7):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Cabanillas ME, de Souza JA, Geyer S, Wirth LJ, Menefee ME, Liu SV, Shah K, Wright J, Shah MH. Cabozantinib As Salvage Therapy for Patients With Tyrosine Kinase Inhibitor-Refractory Differentiated Thyroid Cancer: Results of a Multicenter Phase II International Thyroid Oncology Group Trial. J Clin Oncol. 2017 Oct 10;35(29):3315-3321. doi: 10.1200/JCO.2017.73.0226. Epub 2017 Aug 17. PMID 28817373

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2013 and January 2015 patients were enrolled by ITOG investigators at six centers in the United States.
Groups:
- Treatment (Cabozantinib-s-malate): Patients receive Cabozantinib 60mg PO QD with dose escalation to 80mg QD or dose reduction to 40mg daily or 20mg. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Cabozantinib-s-malate)
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cabozantinib-s-malate)
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 64 [41 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate, Defined as the Proportion of Patients Who Have Had a PR or CR as Assessed by the RECIST Version (v)1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabozantinib-s-malate)
Number analyzed (Participants) | 25
Participants | 10

2. Secondary Outcome: Bone Turnover, as Measured by Serum and Urinary Markers of Bone Turnover
Time Frame: Up to 2 months
Population: Data not collected to be analyzed at this time
Arm/Group | Treatment (Cabozantinib-s-malate)
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Objective Response as Assessed by the RECIST v1.1
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From date of documentation of response to the date of progression or death, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Cabozantinib-s-malate)
Number analyzed (Participants) | 25
months | 11.3 [10.3 to NA] — not evaluable

4. Secondary Outcome: Expression Levels of Predictive Biomarkers of Response by Immunohistochemistry in Archived Tumor Tissue
Description: These baseline levels will be quantitatively summarized and graphically explored, in particular in terms of how they relate to clinical outcomes of interest. Analyses exploring differences in these angiogenic and correlative markers in relation to clinical outcomes will be largely hypothesis-generating. With limited numbers of patients patterns of difference will primarily be looked for using graphical analyses; these can include plots of these marker levels in relation to clinical outcomes to identify potential patterns of interest.
Time Frame: Baseline
Population: Data has not been collected and analyzed at this time
Arm/Group | Treatment (Cabozantinib-s-malate)
Number analyzed (Participants) | 0

5. Secondary Outcome: Genotype of Biomarkers Potentially Predictive of Response
Description: as for outcome 4
Time Frame: Baseline
Population: Data not collected to be analyzed at this time
Arm/Group | Treatment (Cabozantinib-s-malate)
Number analyzed (Participants) | 0

6. Secondary Outcome: Incidence of Severe (Grade 3+) Adverse Events, Graded According to the National Cancer Institute CTCAE v4.0
Description: The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. Tolerability of the regimens will be assessed through assessing the number of patients who required dose modifications and/or dose delays. In addition, the proportion of patients who go off treatment due to adverse reactions or even those who refuse further treatment for lesser toxicities that inhibit their willingness to continue participation on the trial will be captured.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabozantinib-s-malate)
Number analyzed (Participants) | 25
Participants
  Left ventricular systolic dysfunction | 1
  asymptomatic increased lipase | 1
  osteonecrosis of the jaw | 1
  decubitus ulcer | 1
  pneumonia | 1
  meningitis | 1
  perianal hidradenitis suppurativa | 1

7. Secondary Outcome: Overall Survival
Description: The Kaplan-Meier method will be used.
Time Frame: Time from start of treatment to time of death, assessed up to 1 year
Population: the end of the range was not reached
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Cabozantinib-s-malate)
Number analyzed (Participants) | 25
months | 34.7 [18.3 to NA] — Not reached

8. Secondary Outcome: Percent Change in Serum Tumor Marker Thyroglobulin Levels
Description: Side-by-side boxplots will be used to assess possible differences in this change between responders and non-responders, and scatterplots can assess the influence of baseline thyroglobulin levels on these measures of change.
Time Frame: Baseline to 6 months
Population: Data not collected to be analyzed at this time
Arm/Group | Treatment (Cabozantinib-s-malate)
Number analyzed (Participants) | 0

9. Secondary Outcome: Progression-free Survival
Description: The Kaplan-Meier method will be used.
Time Frame: Time from start of treatment to time of progression or death, whichever occurs first, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Cabozantinib-s-malate)
Number analyzed (Participants) | 25
months | 12.7 [10.9 to 34.7]

10. Secondary Outcome: Response of Cabozantinib-s-malate in Bone Metastasis (Bone Metastasis-specific Progression Free Survival) as Evaluated by Functional Imaging
Time Frame: Up to 2 months
Population: Data not collected to be analyzed at this time
Arm/Group | Treatment (Cabozantinib-s-malate)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The National Cancer Institutes (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 was utilized for Adverse event reporting.
Arm/Group | Treatment (Cabozantinib-s-malate)
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 7/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cabozantinib-s-malate) (N=25)
Thrombotic (Vascular disorders) | 1 (1)
Deep venous thrombosis (Vascular disorders) | 1 (1)
Perianal hidradenitis suppurativa (Skin and subcutaneous tissue disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Asymptomatic increased lipase (Metabolism and nutrition disorders) | 1 (1)
Osteonecrosis of the jaw (Gastrointestinal disorders) | 1 (1)
decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Meningitis (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cabozantinib-s-malate) (N=25)
Fatigue (General disorders) | 19 (19)
Anorexia (Metabolism and nutrition disorders) | 16 (16)
Weight Loss (Investigations) | 15 (15)
Dysgeusia (Nervous system disorders) | 12 (12)
Oral mucositis (Gastrointestinal disorders) | 14 (14)
Dry mouth (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 16 (16)
Vomiting (Gastrointestinal disorders) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 18 (18)
Other GI (Gastrointestinal disorders) | 10 (10)
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 19 (19)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Other dermatologic disorder (Skin and subcutaneous tissue disorders) | 10 (10)
Hypertension (Vascular disorders) | 12 (12)
Proteninuria (Vascular disorders) | 8 (8)
Bleeding (Vascular disorders) | 6 (6)
Pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Headache (Nervous system disorders) | 6 (6)
Other muscoskeletal (Musculoskeletal and connective tissue disorders) | 3 (3)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Peripherial neuropathy (Musculoskeletal and connective tissue disorders) | 3 (3)
Liver transaminase elevation (Metabolism and nutrition disorders) | 20 (20)
Hypomagnesemia (Metabolism and nutrition disorders) | 14 (14)
Lipase or amylase elevation (Metabolism and nutrition disorders) | 7 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 12 (12)
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (9)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 6 (6)
Alkaline phosphatase elevation (Metabolism and nutrition disorders) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Amenia (Blood and lymphatic system disorders) | 9 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8)
Leukopenia (Blood and lymphatic system disorders) | 7 (7)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less